CLINICAL TRIAL: NCT01309321
Title: Development and Evaluation of Perinatal Handwashing Promotion for Improved Maternal Handwashing Behavior
Brief Title: Perinatal Handwashing Intervention in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: State University of New York at Buffalo (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-10036
Record Dates: First submitted 2010-10-07; First posted 2011-03-07 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2010-10

CONDITIONS: Sepsis; Umbilical Cord; Infection
Keywords: Perinatal; Handwashing; Neonatal; Morbidity; Mortality; Primiparous; Health behavior; Developing countries; Sepsis; Omphalitis; Infectious disease; Bangladesh
MeSH Terms: conditions — Sepsis; Infections; Health Behavior; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perinatal Handwashing Intervention Arm (Experimental)
  Interventions: Behavioral: Perinatal Handwashing Promotion
- Neonatal Health Promotion (Active Comparator)
  Interventions: Behavioral: Neonatal Health Promotion

INTERVENTIONS:
Behavioral: Perinatal Handwashing Promotion — Pregnancy may serve as a unique opportunity to improve maternal handwashing behavior more deeply and sustainably than a handwashing promotion intervention at a different time. Primiparous women will receive an intensive handwashing promotion program delivered at 3 in-home visits between one month prenatal and 1 week post natal. The program will promote handwashing benefits, provide hardware to reduce barriers to handwashing, and educate mothers about the critical times for handwashing. Mothers will also receive an essential neonatal care package with information on clean delivery, hypothermia prevention, breastfeeding counseling, umbilical cord care, and identification of neonatal danger signs.
  Arms: Perinatal Handwashing Intervention Arm
Behavioral: Neonatal Health Promotion — Mothers will receive an essential neonatal care package with information on clean delivery, hypothermia prevention, breastfeeding counseling, umbilical cord care, and identification of neonatal danger signs.
  Arms: Neonatal Health Promotion

SUMMARY:
The purpose of this study is to determine if an intensive handwashing intervention administered to primiparous women during their pregnancy can increase maternal handwashing with soap at critical times.

DETAILED DESCRIPTION:
In high neonatal mortality settings, about half of neonatal deaths are estimated to occur because of infectious syndromes such as sepsis, acute respiratory infection, neonatal tetanus, and diarrhea. Promoting handwashing to mothers in the post-neonatal period has been shown to reduce the risk of pneumonia and diarrhea among infants > 28 days old but there is little information on the protective effect of handwashing for neonatal health outcomes. The proposed study will assess motivators and barriers to handwashing with soap among new mothers, and develop and test a hand cleansing promotion intervention in rural Bangladesh. The handwashing behavior change intervention will include approaches to enhance maternal expectations of being a good nurturer, as well as enhancing maternal self-efficacy to carry out handwashing behavior.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women who plan to remain in the study area up to 1 months after birth

Exclusion Criteria:

* Prior live birth

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proportion of critical events where neonatal caregivers wash their hands with soap as a measure of behavior change. | 1 month post-natal
Proportion of critical events where neonatal caregivers wash their hands with soap as a measure of behavior change. | 3 months post-natal
Daily reduction in household soap weight. | 2 weeks post-natal.
Daily reduction in household soap weight. | 1 month post-natal

SECONDARY OUTCOMES:
Incidence density of suspected sepsis in neonates | 1 month post natal
Incidence density of suspected omphalitis in neonates | 1 month post-natal
All cause neonatal mortality rate. | 1 month post-natal.

CONTACTS AND LOCATIONS:
Overall Officials: Sharifa Nasreen, MBBS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; Pavani K. Ram, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- ICDDR,B, Matlab, Bangladesh